CLINICAL TRIAL: NCT07339306
Title: A Novel Fluorescent Ductal Needle With Controllable Detachment for Realtime Localization and Sampling of Micro Lesions in Breast Ducts: a Prospective, Multicenter Study
Brief Title: A Novel Fluorescent Ductal Needle for Localization and Sampling of Micro Lesions in Breast Ducts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, JIAN WEN, Director of the Ninth General Surgery Department, The Fourth Affiliated Hospital of China Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FourthAHChinaMU-PMS
Record Dates: First submitted 2025-12-22; First posted 2026-01-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Mammary Tumor; Nipple Discharge; Breast Ductal Carcinoma In Situ
Keywords: micro lesions; breast duct; fluorescent ductal needle; localization needle; controllable detachment
MeSH Terms: conditions — Breast Neoplasms; Galactorrhea; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Intervention Model Description: Experimental Group: Patients received breast ductal excision surgery utilizing a novel fluorescent localization marker needle.
  Control Group: Patients received breast ductal excision surgery utilizing conventional localization methods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluorescent Localization Group (Experimental): Patients received breast ductal excision surgery utilizing a novel fluorescent localization marker needle.
  Interventions: Device: novel fluorescent localization marker needle
- Conventional Localization Group (Active Comparator): Patients received breast ductal excision surgery utilizing conventional localization methods.
  Interventions: Device: conventional localization marker needle

INTERVENTIONS:
Device: novel fluorescent localization marker needle — novel fluorescent localization needle, which features a controllable shedding quantum dot chiral nanofluorescent coating
  Arms: Fluorescent Localization Group
Device: conventional localization marker needle — conventional localization marker needle, without any coating
  Arms: Conventional Localization Group

SUMMARY:
This prospective, multicenter cohort study investigates the differences in the reliability of rapid pathology compared to postoperative pathology when utilizing a novel fluorescent localization needle equipped with a controllable shedding quantum dot chiral nanofluorescent coating, in contrast to traditional localization techniques for breast duct lesions. The principal objective is to assess the clinical efficacy of this innovative fluorescent localization needle in enabling precise pathological diagnosis of micro lesions in breast ducts.

DETAILED DESCRIPTION:
The diameter of breast ducts is less than 0.7 mm, presenting a significant technical challenge for the precise localization of early-stage, small lesions during surgical and pathological sampling. These early microlesions typically measure only a few millimeters, necessitating surgeons to increase excision margins to minimize the risk of overlooking them. However, this approach complicates the pathologists' ability to accurately identify these microlesions during diagnosis, thereby increasing the likelihood of missed diagnoses and the potential need for additional surgical interventions. Current localization methods, including liquid methylene blue and conventional localization needles, exhibit a high rate of pathological missed diagnoses due to localization inaccuracies and specimen contamination. Consequently, there is an urgent need to develop innovative localization technologies capable of facilitating the precise identification of millimeter-scale microlesions within breast ducts. A prospective multicenter study is required to compare the consistency of intraoperative and postoperative pathological assessments between a novel fluorescent localization needle-featuring a controllable shedding quantum dot chiral nanofluorescent coating-and traditional localization techniques employed in breast duct lesion surgeries. The primary objective is to evaluate the clinical efficacy of this new fluorescent localization needle in enhancing the accuracy of pathological diagnosis of microlesions within breast ducts and to improve the precision of pathological evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-75 years.
2. Patients scheduled to undergo duct excision surgery.
3. Patients who are capable of providing written informed consent and adhering to the study protocols.

Exclusion Criteria:

1. Pregnant or breastfeeding.
2. Patients who have known allergy to quantum-dot materials or localization needle components.
3. Patients with active hepatitis B or C infection with detectable viral load.
4. Patients with unstable cardiovascular disease (e.g., recent myocardial infarction, uncontrolled arrhythmia, NYHA class III-IV heart failure).
5. Patients with history of neurological or psychiatric disorders that may impair compliance (e.g., epilepsy, dementia).
6. Patients who concurrent participation in another interventional clinical trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
pathological assessment concordance rates | From enrollment to the end of treatment at 6 weeks
  Evaluate and compare the discrepancies in the consistency of intraoperative frozen and postoperative paraffin-embedded pathological assessments between subjects undergoing breast duct excision surgery utilizing a novel fluorescent localization marker needle and those employing conventional localization methods.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Wen, MD, Principal Investigator — The Fourth Affiliated Hospital of China Medical University
Locations (1):
- The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No